CLINICAL TRIAL: NCT01803672
Title: Effectiveness of an Integrated Adventure-Based Training and Health Education Programme in Promoting the Adoption and Maintenance of Regular Physical Activity Among Childhood Cancer Survivors
Brief Title: Effectiveness of an Integrated Programme in Promoting the Regular Physical Activity Among Childhood Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 102009189
Record Dates: First submitted 2013-02-26; First posted 2013-03-04 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: Malignant Childhood Neoplasm
Keywords: Adventure-Based training; Health education; childhood cancer; physical activity
MeSH Terms: conditions — Neoplasms; Health Education; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- health talk and adventure-based training (Experimental): Participate will join a four-day integrated health education and adventure-based training programme, which contains education talks, workshop and adventure-based training activities. The programme will be implemented on four different days within six months in a day camp training centre. The integrated programme will be implemented in small group with maximum 15 participants in one group. Health education talks and workshop will be implemented in between adventure-based training activities in day camp centre, which will be conducted by healthcare professionals working in a local university.
  Interventions: Behavioral: health talk and adventure-based training
- Placebo Control (Placebo Comparator): Participants will receive an amount of time and attention that mimicked that received by the experimental group, but which is thought not to have any specific effect on the outcome measures. They will be invited to attend leisure activities organized by a community centre in four different days during the study period. Activities will include cartoon film shows, handicraft workshops, chess games, health talks on the prevention of influenza and healthy diet, day visit to museum and theme park.
  Interventions: Behavioral: Placebo control

INTERVENTIONS:
Behavioral: health talk and adventure-based training — To develop an integrated programme for Hong Kong Chinese childhood cancer survivors, an advisory committee was set up which included the three healthcare professionals (researchers), two school principals, two professional adventure-based trainers and one assistant professor of Sports and Recreation Management, ensuring the adequate 'dosage' of the intervention and the feasibility of implementing such programme for Hong Kong childhood cancer surviviors.
  Arms: health talk and adventure-based training
Behavioral: Placebo control — They will be invited to attend leisure activities organized by a community centre in four different days during the study period. Activities will include cartoon film shows, handicraft workshops, chess games, health talks on the prevention of influenza and healthy diet, day visit to museum and theme park.
  Arms: Placebo Control

SUMMARY:
Background.There is some evidence that engaging in regular moderate-intensity physical activity may help ameliorate cancer-related fatigue experienced by childhood cancer survivors, which eventually improve their quality of life. Nevertheless, there is growing concern about declining levels of physical activity in childhood cancer survivors.

Purposes. To examine the effectiveness of an integrated adventure-based training and health education programme in promoting the adoption and maintenance of regular physical activity, reducing fatigue and improving the quality of life among Hong Kong Chinese childhood cancer survivors.

Design and Subjects. A randomised controlled trial (RCT), two-group pre-test and repeated post-test, between subjects design was conducted. Recruitment of subjects was carried out through the Sunshine Parents Club, which is a non-profit voluntary organization with the aim to provide education and psychological support to parents of Hong Kong Chinese childhood cancer survivors.

Intervention. Participants in the placebo control group received an amount of time and attention (leisure activities organized by a community centre) that mimicked that received by the experimental group. Participants in the experimental group joined a four-day integrated adventure-based training and health education programme, which contained education talks, a workshop and adventure-based training activities.

DETAILED DESCRIPTION:
The aim of this study was to examine the effectiveness of an integrated adventure-based training and health education programme in promoting the exercise behavior changes, enhancing the physical activity levels, self-efficacy, reducing fatigue and improving the quality of life of Hong Kong Chinese childhood cancer survivors.

Intervention

Placebo control group

Participants received medical follow-up according to the schedule of the oncology units. Besides, participants received an amount of time and attention that mimicked that received by the experimental group, but which is thought not to have any specific effect on the outcome measures. They were invited to attend leisure activities organized by a community centre in four different days during the study period. Activities included cartoon film shows, handicraft workshops, chess games, health talks on the prevention of influenza and healthy diet, day visit to museum and theme park.

Experimental group

Besides receiving medical follow-up, participants joined a four-day integrated adventure-based training and health education programme, which contains education talks, a workshop to work out a feasible individual action plan for regular physical activity and adventure-based training activities. Previous research showed that working out individual action plan is important, which can increase the possibility for people to turn their intentions into health promotion action. The content of the education talks were tailor-made for participants in which they did not engage in regular physical activity.

To ensure the dosage of intervention delivered in terms of the amount, frequency, duration, and breadth would be adequate to assess the quality and to manage outcomes, such as physical activity levels, self-efficacy, stages of change and quality of life, the following measures were taken. An advisory committee was set up with the purpose to develop an appropriate integrated programme for Hong Kong Chinese childhood cancer survivors. The committee included the researcher, an assistant professor at a local university with considerable experience of conducting psychological interventions among children, a paediatric oncologist and a oncology nurse specialist with rich experience in taking care of children with cancer, two professional adventure-based trainers and one assistant professor of Sports and Recreation Management with extensive experience and professional knowledge in conducting adventure-based training for children. In addition, the content of the programme that related to adventure-based training activities was sent to a professional adventure-based training centre for content validation. The programme was implemented on four different days within six months in a day camp training centre, such as at 2-week, 2-month, 4-month and 6-month after the day of recruitment. The programme was implemented in small group with maximum 12 participants in one group. Health education talks and workshop were implemented in between adventure-based training activities in day camp centre, which were conducted by healthcare professionals working in a local university. Adventure-based training activities were led by two qualified adventure-based training instructors with extensive experience and professional knowledge in conducting such training for children. Additionally, at least two healthcare professionals joined the adventure-based training to monitor the physical condition of the survivors and their fitness to join the adventure-based training activities.

Data Collection Methods

Data Collection Methods Approval for the study was obtained from the hospital ethics committees. To identify potential subjects, a leaflet containing details of the study and a demographic sheet have been mailed to all parents of childhood cancer survivors in the Sunshine Parents Club. If children and their parents are interested in the research, they can return the demographic sheet by using the enclosed return-envelop to convey their willingness to participate in the study. A briefing session will then be conducted in the out-patient clinic to those eligible children and parents. Written consent has been obtained from the parents after they were told the purposes of the study, although they were of course given the option of allowing or refusing the involvement of their child. The children has also been invited to put their names on a special children's assent form and told that their participation is voluntary.

After obtaining demographic data of participants, they have been asked to respond to the Chinese version of the FS-C/FS-A, PA-SE, CUHK-PARCY, PASCQ and PedsQL. They have also been assessed for muscle strength using a hand-held dynamometer. Participants have been randomly assigned to the experimental and control groups. All participants received a telephone call inviting them to join the interventions according to their group assignment at an appointed time. Data collection has been conducted again at 3, 6, 9 and 12 months after starting the intervention. All participants has been informed that there would be home visits for data collection.

Analysis

The Statistical Package for Social Sciences (SPSS) software, version 19.0 for Windows will be used to analyze quantitative data. Intention-to-treat analysis will be used and missing data will be substituted by the last-observation-carried-forward procedure. The comparability of the experimental and control groups will be assessed by using inferential statistics (independent t-test and chi-squared test). Descriptive statistics will be used to calculate the mean scores and standard deviation of different scales. Mixed between-within subjects ANOVA (split-plot ANOVA) will be used to determine whether the adventure-based training programme was effective in reducing fatigue, increasing childhood cancer survivors' levels of physical activity, self-efficacy and muscle strength and enhancing their quality of life. In addition, Friedman Test will be used to determine any changes in stages of change between the experimental and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong Chinese childhood cancer survivors defined here as having completed treatment at least six months previously
* between 7 and 18 years of age
* able to speak Cantonese and read Chinese
* did not engage in regular physical activity for the past 6 months

Exclusion Criteria:

* childhood cancer survivors with evidence of recurrence or second malignancies
* those with physical impairment or cognitive and learning problems identified from their medical records

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 71 (Actual)
Dates: Start 2012-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
change in levels of cancer-related fatigue from baseline at 6-month follow-up between intervention and control group | 6-month follow-up
  The primary outcomes are levels of cancer-related fatigue at 6 months after starting the intervention among the two groups. The Fatigue Scale - Child will be used to assess the fatigue of subjects who are 7 to 12 years old. For those aged 13 to 18, their fatigue levels will be measured by the Fatigue Scale - Adolescent.

SECONDARY OUTCOMES:
change in levels of cancer-related fatigue from baseline at 3-month follow-up between intervention and control group | 3-month follow-up
  The Fatigue Scale - Child will be used to assess the fatigue of subjects who are 7 to 12 years old. For those aged 13 to 18, their fatigue levels will be measured by the Fatigue Scale - Adolescent.
change in levels of cancer-related fatigue from baseline at 9-month follow-up between intervention and control group | 9-month follow-up
  The Fatigue Scale - Child will be used to assess the fatigue of subjects who are 7 to 12 years old. For those aged 13 to 18, their fatigue levels will be measured by the Fatigue Scale - Adolescent.
change in levels of cancer-related fatigue from baseline at 12-month follow-up between intervention and control group | 12-months follow-up
  The Fatigue Scale - Child will be used to assess the fatigue of subjects who are 7 to 12 years old. For those aged 13 to 18, their fatigue levels will be measured by the Fatigue Scale - Adolescent.
levels of cancer-related fatigue at Baseline | Baseline
  The Fatigue Scale - Child will be used to assess the fatigue of subjects who are 7 to 12 years old. For those aged 13 to 18, their fatigue levels will be measured by the Fatigue Scale - Adolescent.
change in physical activity levels from baseline at 6-month follow-up between intervention and control group | 6-month follow-up
  The physical activity levels of participants will be assessed using the CUHK-PARCY, which is an 11-item activity rating modified from the Jackson Activity Coding and the Godin-Shephard Activity Questionnaire Modified for Adolescents. Participant will be asked to respond to the Chinese version of the CUHK-PARCY at 6 months after starting the intervention.
change in physical activity levels from baseline at 3-month follow-up between intervention and control group | 3-month follow-up
  The physical activity levels of participants will be assessed using the CUHK-PARCY, which is an 11-item activity rating modified from the Jackson Activity Coding and the Godin-Shephard Activity Questionnaire Modified for Adolescents. Participant will be asked to respond to the Chinese version of the CUHK-PARCY at 6 months after starting the intervention.
change in physical activity levels from baseline at 9-month follow-up between intervention and control group | 9-month follow-up
  The physical activity levels of participants will be assessed using the CUHK-PARCY, which is an 11-item activity rating modified from the Jackson Activity Coding and the Godin-Shephard Activity Questionnaire Modified for Adolescents. Participant will be asked to respond to the Chinese version of the CUHK-PARCY at 9 months after starting the intervention.
change in physical activity levels from baseline at 12-month follow-up between intervention and control group | 12-month follow-up
  The physical activity levels of participants will be assessed using the CUHK-PARCY, which is an 11-item activity rating modified from the Jackson Activity Coding and the Godin-Shephard Activity Questionnaire Modified for Adolescents. Participant will be asked to respond to the Chinese version of the CUHK-PARCY at 12 months after starting the intervention.
Physical activity levels activity at Baseline | Baseline
  The physical activity levels of participants will be assessed using the CUHK-PARCY, which is an 11-item activity rating modified from the Jackson Activity Coding and the Godin-Shephard Activity Questionnaire Modified for Adolescents. Participants will be asked to respond to the Chinese version of the CUHK-PARCY before randomization.
Stages of Change at baseline | Baseline
  The current stages of exercising patterns for participants will be evaluated by an adapted version of PASCQ. It is a binary type (yes/no) questionnaire, and contains four items. Participants will answer each question about their physical activity practices with a 'yes' or a 'no'. According to these responses, they will be classified into five different stages by means of a scoring algorithm. Participant will be asked to respond to the Chinese version of the PASCQ before the randomization.
change in stages of change from baseline at 3-month follow-up between intervention and control group | 3-month follow up
  The current stages of exercising patterns for participants will be evaluated by an adapted version of PASCQ. It is a binary type (yes/no) questionnaire, and contains four items. Participants will answer each question about their physical activity practices with a 'yes' or a 'no'. According to these responses, they will be classified into five different stages by means of a scoring algorithm. Participant will be asked to respond to the Chinese version of the PASCQ 3 months after starting the intervention.
change in stages of change from baseline at 6-month follow-up between intervention and control group | 6-month follow up
  The current stages of exercising patterns for participants will be evaluated by an adapted version of PASCQ. It is a binary type (yes/no) questionnaire, and contains four items. Participants will answer each question about their physical activity practices with a 'yes' or a 'no'. According to these responses, they will be classified into five different stages by means of a scoring algorithm. Participant will be asked to respond to the Chinese version of the PASCQ 6 months after starting the intervention.
change in stages of change from baseline at 9-month follow-up between intervention and control group | 9-month follow up
  The current stages of exercising patterns for participants will be evaluated by an adapted version of PASCQ. It is a binary type (yes/no) questionnaire, and contains four items. Participants will answer each question about their physical activity practices with a 'yes' or a 'no'. According to these responses, they will be classified into five different stages by means of a scoring algorithm. Participant will be asked to respond to the Chinese version of the PASCQ 9 months after starting the intervention.
change in stages of change from baseline at 12-month follow-up between intervention and control group | 12-month follow up
  The current stages of exercising patterns for participants will be evaluated by an adapted version of PASCQ. It is a binary type (yes/no) questionnaire, and contains four items. Participants will answer each question about their physical activity practices with a 'yes' or a 'no'. According to these responses, they will be classified into five different stages by means of a scoring algorithm. Participant will be asked to respond to the Chinese version of the PASCQ 12 months after starting the intervention.
physical activity self-efficacy at baseline | baseline
  The PA-SE will be used to measure the children's self-confidence in their ability to participate in various age-appropriate physical activities. The PA-SE includes five items in which children are asked if they are 'not sure', 'a little sure' or 'very sure' that they can do such things such as 'keep up a steady pace without stopping for 15-20 min'. Higher scores indicate higher self-efficacy. Participants will be asked to respond to the Chinese version of the PA-SE before the randomization.
change in physical activity self-efficacy from baseline at 3-month follow-up between intervention and control group | 3-month follow up
  The PA-SE will be used to measure the children's self-confidence in their ability to participate in various age-appropriate physical activities. The PA-SE includes five items in which children are asked if they are 'not sure', 'a little sure' or 'very sure' that they can do such things such as 'keep up a steady pace without stopping for 15-20 min'. Higher scores indicate higher self-efficacy. Participants will be asked to respond to the Chinese version of the PA-SE 3 months after starting the intervention.
change in physical activity self-efficacy from baseline at 6-month follow-up between intervention and control group | 6-month follow up
  The PA-SE will be used to measure the children's self-confidence in their ability to participate in various age-appropriate physical activities. The PA-SE includes five items in which children are asked if they are 'not sure', 'a little sure' or 'very sure' that they can do such things such as 'keep up a steady pace without stopping for 15-20 min'. Higher scores indicate higher self-efficacy. Participants will be asked to respond to the Chinese version of the PA-SE 6 months after starting the intervention.
change in physical activity self-efficacy from baseline at 9-month follow-up between intervention and control group | 9-month follow up
  The PA-SE will be used to measure the children's self-confidence in their ability to participate in various age-appropriate physical activities. The PA-SE includes five items in which children are asked if they are 'not sure', 'a little sure' or 'very sure' that they can do such things such as 'keep up a steady pace without stopping for 15-20 min'. Higher scores indicate higher self-efficacy. Participants will be asked to respond to the Chinese version of the PA-SE 9 months after starting the intervention.
change in physical activity self-efficacy from baseline at 12-month follow-up between intervention and control group | 12-month follow up
  The PA-SE will be used to measure the children's self-confidence in their ability to participate in various age-appropriate physical activities. The PA-SE includes five items in which children are asked if they are 'not sure', 'a little sure' or 'very sure' that they can do such things such as 'keep up a steady pace without stopping for 15-20 min'. Higher scores indicate higher self-efficacy. Participants will be asked to respond to the Chinese version of the PA-SE 12 months after starting the intervention.
quality of life at baseline | baseline
  The PedsQL will be used to measure quality of life among childhood cancer survivors. The instrument comprises 23 items grouped into four subscales: physical functioning (8 items), emotional functioning (5 items), social functioning (5 items) and school functioning (5 items). Participants will be asked how much of a problem has been experienced over the last month, with rating from 0 to 4. Higher scores indicate better quality of life. Participant will be asked to respond to the Chinese version of the PedsQL before the randomization.
change in quality of life from baseline at 3-month follow-up between intervention and control group | 3-month follow up
  The PedsQL will be used to measure quality of life among childhood cancer survivors. The instrument comprises 23 items grouped into four subscales: physical functioning (8 items), emotional functioning (5 items), social functioning (5 items) and school functioning (5 items). Participants will be asked how much of a problem has been experienced over the last month, with rating from 0 to 4. Higher scores indicate better quality of life. Participant will be asked to respond to the Chinese version of the PedsQL 3 months after starting the intervention.
change in quality of life from baseline at 6-month follow-up between intervention and control group | 6-month follow up
  The PedsQL will be used to measure quality of life among childhood cancer survivors. The instrument comprises 23 items grouped into four subscales: physical functioning (8 items), emotional functioning (5 items), social functioning (5 items) and school functioning (5 items). Participants will be asked how much of a problem has been experienced over the last month, with rating from 0 to 4. Higher scores indicate better quality of life. Participant will be asked to respond to the Chinese version of the PedsQL 6 months after starting the intervention.
change in quality of life from baseline at 9-month follow-up between intervention and control group | 9-month follow up
  The PedsQL will be used to measure quality of life among childhood cancer survivors. The instrument comprises 23 items grouped into four subscales: physical functioning (8 items), emotional functioning (5 items), social functioning (5 items) and school functioning (5 items). Participants will be asked how much of a problem has been experienced over the last month, with rating from 0 to 4. Higher scores indicate better quality of life. Participant will be asked to respond to the Chinese version of the PedsQL 9 months after starting the intervention.
change in quality of life from baseline at 12-month follow-up between intervention and control group | 12-month follow up
  The PedsQL will be used to measure quality of life among childhood cancer survivors. The instrument comprises 23 items grouped into four subscales: physical functioning (8 items), emotional functioning (5 items), social functioning (5 items) and school functioning (5 items). Participants will be asked how much of a problem has been experienced over the last month, with rating from 0 to 4. Higher scores indicate better quality of life. Participant will be asked to respond to the Chinese version of the PedsQL 12 months after starting the intervention.
muscle strength at baseline | baseline
  the isokinetic strength of muscles will be measured by a dynamometer using a break and make technique before randomization.
change in muscle strength from baseline at 3-month follow-up between intervention and control group | 3-month follow up
  The isokinetic strength of muscles will be measured by a dynamometer using a break and make technique 3 months after starting the intervention.
change in muscle strength from baseline at 6-month follow-up between intervention and control group | 6-month follow up
  The isokinetic strength of muscles will be measured by a dynamometer using a break and make technique 6 months after starting the intervention.
change in muscle strength from baseline at 9-month follow-up between intervention and control group | 9-month follow up
  The isokinetic strength of muscles will be measured by a dynamometer using a break and make technique 9 months after starting the intervention.
change in muscle strength from baseline at 12-month follow-up between intervention and control group | 12-month follow up
  The isokinetic strength of muscles will be measured by a dynamometer using a break and make technique 12 months after starting the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: William Ho Cheung Li, PhD, Principal Investigator — The School of Nursing, The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No